CLINICAL TRIAL: NCT00414869
Title: Preliminary Efficacy And Tolerability Of Oral NCX-1000 After Repeated Administrations In Patients With Portal Hypertension: A Double-Blind Dose Escalating Study
Brief Title: Preliminary Efficacy and Tolerability of NCX-1000 After Repeated Oral Doses in Patients With Elevated Portal Pressure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary analysis of 11 patients did not demonstrate the efficacy required.
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCXDE05-02
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Portal Hypertension
Keywords: Liver; Portal pressure; Fibrosis; Nitric oxide
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — 2-methyl-3-(2-((4-nitrooxybutyloxy)carbonyl)vinyl)phenyl ursodeoxycholic acid ester

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NCX-1000 (Experimental): Experimental drug under evaluation
  Interventions: Drug: NCX-1000
- Placebo (Placebo Comparator): Placebo powder
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NCX-1000 — 500 mg powder sachets to be taken as 1, 2, or 4 sachets twice daily, PO x 16 days
  Arms: NCX-1000
Drug: Placebo — Inactive powder matching NCX-1000
  Arms: Placebo

SUMMARY:
Chronic liver diseases are often characterized by portal hypertension, a major complication involving haemodynamic changes due to increased intrahepatic vascular resistance. It has become well established that nitric oxide (NO) plays a crucial role in the haemodynamic abnormalities that develop in chronic portal hypertension.

NCX-1000 is a NO-releasing derivative of ursodeoxycholic acid that would compensate for the defective liver NO production in cirrhosis.

This study intends to demonstrate the desired therapeutic activity (reduction in portal pressure) in a small number of target patients, to assess the safety and tolerability after repeated oral administrations of NCX-1000, and to get preliminary pharmacokinetic data in this population.

DETAILED DESCRIPTION:
Brief summary is complete. Study is closed.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patients of at least 18 years old
* HVPG > 12 mm Hg in fasting state on Day 1
* Free of any other condition (except liver failure) that may alter absorption, distribution, or elimination of drugs

Exclusion Criteria:

* Oesophageal bleeding in the previous 30 days
* Known intolerance to ursodeoxycholic acid or nitrates
* Liver cancer or liver metastasis from another cancer
* Portal hypertension secondary to venous thrombosis
* Presence of Transjugular Intrahepatic Portosystemic Shunt (TIPS)
* Severe liver failure (Child-Pugh C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The Hepatic Venous Pressure Gradient (HVPG) will be evaluated at entry (Day 1) and after the Maximal Tolerated Dose (MTD) on Day 16, in fasting and post-prandial (after a standardized liquid breakfast) states. | Day1 and Day 16
  The portal pressure, as determined by HVPG, was obtained by subtracting the free hepatic venous pressure from the wedged hepatic venous pressure and rounded to the nearest 0.5 or integer value.The pressures were recorded 3 times for each evaluation and the HVPG value was the mean of the 3 Recordings

SECONDARY OUTCOMES:
Safety parameters: systolic and diastolic blood pressures, heart rate, physical examination, laboratory tests and Adverse Events (AEs) | At various times
  Usual safety parameters. Blood pressures were assessed every 30 minutes for 4 hours after drug intake. Other parameters were assessed or reported at Study visits
Plasma levels of NCX-1000 and its main metabolites will be evaluated to get preliminary pharmacokinetic data. | 0, 1, 2, 3, and 4 hours after the first 3 doses anf after the last dose
  Usual pharmacokinetic (PK) evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Bosch, MD, Principal Investigator — Clinic Barcelona Hospital Universatiri
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain